CLINICAL TRIAL: NCT01683188
Title: A Multi-Center Study of High Dose Aldesleukin (Interleukin-2) + Vemurafenib Therapy in Patients With BRAFV600 Mutation Positive Metastatic Melanoma
Brief Title: HD IL-2 + Vemurafenib in Patients With BRAF Mutation Positive Metastatic Melanoma
Acronym: PROCLIVITY01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow accrual led to early closure.
Sponsor: Clinigen, Inc. (Industry)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12PLK01
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; skin cancer; Stage IV
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Vemurafenib; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Other): Patients who have received less than 7 weeks vemurafenib dosing prior to treatment with HD IL-2
  Interventions: Drug: vemurafenib + HD IL-2
- Cohort 2 (Other): Patients who have receive >7 weeks to 18 weeks vemurafenib dosing prior to treatment with HD IL-2
  Interventions: Drug: vemurafenib + HD IL-2

INTERVENTIONS:
Drug: vemurafenib + HD IL-2
  Other Names: Proleukin

SUMMARY:
This is a research study to evaluate treatment of metastatic melanoma patients with a combination of drugs. The combination being studied is vemurafenib (also known as Zelboraf®) and High Dose Interleukin-2 (abbreviated as HD IL-2 and known as Proleukin®). The combination of vemurafenib and HD IL-2 immunotherapy may enhance the response.

DETAILED DESCRIPTION:
This will be an open-label, uncontrolled two-arm, multi-center study in patients with metastatic melanoma with BRAFV600 oncogene mutations. Patients will initially receive treatment with vemurafenib interspersed with two courses of High Dose IL-2 (HD IL-2). Patients are eligible for the study if they have melanoma positive for the BRAFV600 mutation, have been on vemurafenib therapy for 0-18 weeks, have responding or stable disease if on vemurafenib, and meet the requirements for dosing with HD IL-2 and all protocol inclusion and exclusion criteria.

Two Cohorts will be enrolled, differing only in how they are characterized prior to HD IL-2 treatment:

Cohort 1: will consist of 135 patients naïve to vemurafenib and HD IL-2 therapy. Patients in Cohort 1 will have an initial evaluation and receive a defined 6 (± 1) week course of vemurafenib before beginning HD IL-2. This Cohort will be used to define study size and statistical validity with the comparator being historic controls (using data from the BRAF positive patients from the Melanoma SELECT study Protocol IIT10PLK06).

Cohort 2: will consist of up to 50 patients who have been on vemurafenib therapy for >7 to 18 weeks with stable or responding disease before starting HD IL-2. Patients in Cohort 2 will have an initial evaluation and will begin HD IL-2 treatment after >7 to 18 weeks of treatment with vemurafenib. This Cohort is designed to evaluate whether additive or synergistic clinical benefit or toxicity is observed in BRAFV600 mutation positive metastatic melanoma patients treated with vemurafenib as a single agent for >7 to18 weeks prior to the first course of HD IL-2 therapy in conjunction with continued vemurafenib.

Patients in both cohorts will discontinue dosing vemurafenib prior to each treatment with HD IL-2 and resume dosing after each discharge. Patients will receive up to two courses (four cycles) of HD IL-2 and will be evaluated for their disease responses at 10 weeks (±3 weeks) from the start of HD IL-2 dosing, and 26 weeks (±3 weeks) from the start of HD IL-2 dosing. QTc intervals will be reviewed daily for changes during each cycle of HD IL-2 dosing.

Administration of vemurafenib and HD IL-2 will be according to the respective Package Inserts and according to the Institution's standard of care. The investigator will determine the number of HD IL-2 cycles each patient will receive, according to the investigator's discretion and medical judgment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older.
* Confirmed and measurable metastatic melanoma with the BRAFV600 mutation.
* Patients with at least one metastatic melanoma lesion accessible. for biopsy prior to vemurafenib treatment if no archived tissue is available.
* Meet the requirements for HD IL-2 therapy per institutional guidelines.
* Meet the requirements for vemurafenib therapy per institutional guidelines.
* Patient must be willing to provide written Informed Consent and participate in study procedures as described in the 12PLK01. Patients consented for 12PLK01 will also be asked to participate in the 10PLK13 PROCLAIM (Proleukin®) registry study.

Exclusion Criteria:

* A patient will not be considered eligible for study participation if any of the following exclusion criteria are met:
* Prior therapy of metastatic disease with any of the following: IL-2, Ipilimumab, or other highly selective BRAF, MEK, NRAS, cMET inhibitors (e.g. GSK2118436 or GSK1120212) and TKIs.

  * Exception: with a 6 week washout the following are allowed:

    * Adjuvant Ipilimumab,
    * Anti PD-1, Anti PD L-1
* Exclusion for Cohort 1 only: vemurafenib treatment >7 weeks.
* Exclusion for Cohort 2 only: vemurafenib treatment <7 weeks. (eligible for Cohort 1) or >18 weeks.
* QTc interval of >500ms.
* Patients with known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) or other infectious hepatitis.
* Pregnant, nursing or planning to become pregnant.
* Untreated brain metastases. (Brain metastases that have been treated, which no longer require corticosteroid therapy and are without progression by MRI assessment at least 6 weeks after definitive therapy are acceptable.)
* Received investigational drug within 30 days prior to study dosing. Patients may participate in non-interventional or observational clinical study (ies)
* Concomitant disease or condition that would interfere with the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assess Complete Response (CR) rate in BRAFV600 mutation positive metastatic melanoma patients who have received vemurafenib plus HD IL-2 at 10 (±3) weeks from the start of HD IL-2 dosing to assess initial response and 26 (±3) weeks to assess and change | 10 weeks, 26 weeks
  assessment of tumor response in patients with CR or near CR (> 90%) after discontinuation of vemurafenib, based on RECIST criteria
compare safety between patients treated with vemurafenib and HD IL-2 versus historical HD IL-2 alone | through study completion, an average of 1 year
  incidence of adverse events

SECONDARY OUTCOMES:
Compare PFS | 1 year
  compare progression free survival (PFS) from initiation of vemurafenib between Cohort 1 and Cohort 2 patients, compare overall PFS with the historical data using vemurafenib or HD IL-2 alone,

CONTACTS AND LOCATIONS:
Overall Officials: Tharak Rao, MD, Principal Investigator — Prometheus Laboratories
Locations (21):
- United States (21):
  - University Arizona Cancer Center, Tucson, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - MSMC Research Program, Miami Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Loyola University Medical Center, Div of Hematology/Oncology, Maywood, Illinois
  - Luther General Cancer Care Institute, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Hematology/Oncology Clinic, Baton Rouge, Louisiana
  - University of Michigan, Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Providence Cancer Center, Portland, Oregon
  - St. Luke's Hospital, Anderson Campus, Easton, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark JI, Singh J, Ernstoff MS, Lao CD, Flaherty LE, Logan TF, Curti B, Agarwala SS, Taback B, Cranmer L, Lutzky J, Luna TL, Aung S, Lawson DH. A multi-center phase II study of high dose interleukin-2 sequenced with vemurafenib in patients with BRAF-V600 mutation positive metastatic melanoma. J Immunother Cancer. 2018 Jul 27;6(1):76. doi: 10.1186/s40425-018-0387-x. PMID 30053905